CLINICAL TRIAL: NCT03065777
Title: Evaluation of Postoperative Pain After Single Visit Root Canal Treatment Associated With The Three Rotary Systems; ONE ENDO, F6 SkyTper and ProTaper Universal. (Randomized Controlled Clinical Trial)
Brief Title: Postoperative Pain Associated With Three Endodontic Rotary Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola Adel Hassan Hafez, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-11-173
Record Dates: First submitted 2017-02-15; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Acute Pulpitis
Keywords: single file.; ONE ENDO.; F6 SkyTaper.; ProTaper Universal.; irreversible pulpitis.; postoperative pain.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ONE ENDO (Experimental): Single file rotary system
  Interventions: Device: ONE ENDO
- F6 SKYTaper (Experimental): Single file rotary system
  Interventions: Device: F6 SKYTaper
- ProTaper Universal (Active Comparator): Muti-file rotary system
  Interventions: Device: ProTaper Universal

INTERVENTIONS:
Device: ONE ENDO — single file rotary system
  Arms: ONE ENDO
Device: F6 SKYTaper — single file rotary system
  Arms: F6 SKYTaper
Device: ProTaper Universal — multi-file rotary system
  Arms: ProTaper Universal

SUMMARY:
Assessment of postoperative pain after root canal treatment using different rotary systems.

DETAILED DESCRIPTION:
Randomized controlled clinical trial comparing three types of endodontic rotary files to assess their effect on postoperative pain after single visit root canal treatment of premolar teeth diagnosed with acute irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* Systematically healthy patients,
* maxillary or mandibular premolar teeth with acute irreversible pulpitis and indicated for conventional endodontic treatment.

Exclusion Criteria:

* Non-vital teeth,
* teeth with apical periodontitis,
* teeth requiring endodontic retreatment,
* root resorption,
* immature / open apex,
* root canals with radiographic evidence of calcification,
* presence of more than one symptomatic tooth in the same quadrant,
* pregnancy,
* medically compromised patients,
* patients receiving medication for chronic pain,
* patients who have taken analgesics in the last 12 hours before treatment.
* teeth that have initial apical size more than 20,
* teeth that could not be treated in a single session,
* if any evidence of extrusion of root filling material noticed radiographically, patient will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | up to 72 hours after endodontic treatment
  Verbal Rating Scale (VRS) with the following scores:
  0. No pain.
  1. Mild pain: any discomfort of any duration that does not require analgesics.
  2. Moderate pain: pain that requires and is relieved with analgesics.
  3. Severe pain: any pain that is not relieved with analgesics.

SECONDARY OUTCOMES:
Number of analgesics consumed | up to 72 hours after endodontic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ola A. Hafez, MD Student, Principal Investigator — Faculty of Oral and Dental Medicine - Cairo University; Alaa El-Din H. Diab, Professor, Study Chair — Faculty of Oral and Dental Medicine - Cairo University; Kareem G. Abd El-Kader, Assistant Professor, Study Director — Faculty of Oral and Dental Medicine - Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No